CLINICAL TRIAL: NCT02830724
Title: A Phase I/II Study Administering Peripheral Blood Lymphocytes Transduced With a CD70-Binding Chimeric Antigen Receptor to Patients With CD70-Expressing Cancers
Brief Title: Administering Peripheral Blood Lymphocytes Transduced With a CD70-Binding Chimeric Antigen Receptor to People With CD70 Expressing Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160131; 16-C-0131
Record Dates: First submitted 2016-07-12; First posted 2016-07-13 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-18

CONDITIONS: Pancreatic Cancer; Renal Cell Cancer; Breast Cancer; Melanoma; Ovarian Cancer
Keywords: Metastatic Solid Cancers; Renal Cell Cancer; Cell Therapy; CAR T-Cells; Immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Renal Cell; Breast Neoplasms; Melanoma; Ovarian Neoplasms | interventions — Cyclophosphamide; fludarabine; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + escalating doses of anti-hCD70 CAR transduced PBL + high-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Biological: Anti-hCD70 CAR transduced PBL
- 2/Phase II (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MTD of anti-hCD70 CAR transduced PBL + high-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Biological: Anti-hCD70 CAR transduced PBL

INTERVENTIONS:
Drug: Cyclophosphamide — For Phase I, Days -7 and -6:
  Dose Level 1: 15 mg/kg/day x 2 days IV Dose Level 2: 15 mg/kg/day x 2 days IV Dose Level 3: 15 mg/kg/day x 2 days IV Dose Level 4: 15 mg/kg/day x 2 days IV Dose Level 5: 30 mg/kg/day x 2 days IV Dose Level 6: 60 mg/kg/day x 2 days IV
  For Phase II, Days -7 and -6:
  60 mg/kg/day x 2 days IV
Drug: Fludarabine — For Phase I, Days -7 to -5:
  Dose Level 1: 25 mg/m(2)/day x 3 days IVPB Dose Level 2: 25 mg/m(2)/day x 3 days IVPB Dose Level 3: 25 mg/m(2)/day x 3 days IVPB Dose Level 4: 25 mg/m(2)/day x 3 days IVPB Dose Level 5: 25 mg/m(2)/day x 5 days IVPB Dose Level 6: 25 mg/m(2)/day x 5 days IVPB
  For Phase II, Days -7 to -3:
  25 mg/m(2)/day x 5 days IVPB
Drug: Aldesleukin — Aldeskeukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 3 days (maximum 9 doses).
Biological: Anti-hCD70 CAR transduced PBL — Day 0: Cells will be infused intravenously on the Patient Care Unit over 20-30 minutes (2-5 days after the last dose of fludarabine).

SUMMARY:
Background:

In a new cancer therapy, researchers take a person s blood, select a certain white blood cell to grow in the lab, and then change the genes of these cells using a virus. The cells are then given back to the person. This is called gene transfer. For this study, researchers will modify the person s white blood cells with anti-CD70.

Objectives:

To see if a gene transfer with anti-CD70 cells can safely shrink tumors and to be certain the treatment is safe.

Eligibility:

Adults age 18 and older diagnosed with cancer that has the CD70-expressing cancer.

Design:

Participants will be screened with medical history, physical exam, scans, and other tests. They may by admitted to the hospital. Leukapheresis will be performed. For this, blood is removed through a needle in the arm. A machine separates the white blood cells. The rest of the blood is returned through a needle in the other arm.

Eligible participants will have an intravenous catheter placed in their upper chest. Over several days, they will get chemotherapy drugs and the anti-CD70 cells. They will recover in the hospital.

Participants will take an antibiotic for 6 months after treatment. They will repeat leukapheresis.

Participants will visit the clinic every 1-3 months for the first year after treatment, every 6 months for the second year, and then as determined by their physician. Follow-up visits will take 1-2 days. At each visit, participants will have lab tests, imaging studies, and a physical exam.

Throughout the study, blood will be taken and participants will have many tests to determine the size and extent of their tumor and the treatment s impact.

DETAILED DESCRIPTION:
Background:

* We generated a chimeric antigen receptor (CAR) that engages CD70 using its natural ligand CD27, as the binding moiety. Transducing peripheral blood lymphocytes (PBL) with this CAR conveys major histocompatibility complex (MHC)-independent recognition of CD70-expressing target cells, which include renal cell carcinoma and other cancers.
* In co-cultures with CD70+ target cells, anti-hCD70 CAR transduced T cells secrete significant amounts of IFN-gamma with high specificity.

Objectives:

Primary objectives:

* Phase I: Determine the safety of administering PBL transduced with anti-hCD70 CAR in concert with preparative lymphodepletion and high dose interleukin-2 (IL-2; aldesleukin).
* Phase II: Determine if anti-hCD70 CAR-transduced PBL can mediate the regression of CD70 expressing tumors.

Eligibility:

* Patients must be/have:

  * Age >= 18 years and <= 72 years
  * Metastatic or unresectable CD70-expressing cancer which has progressed after standard therapy
* Patients may not have:

  * Allergies or hypersensitivities to high-dose aldesleukin, cyclophosphamide, or fludarabine.

Design:

* This is a phase I/II, single center study of PBL transduced with anti-hCD70 CAR in patients with measurable, unresectable cancer expressing CD70.
* PBMC obtained by leukapheresis will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of these cells to retroviral vector supernatant containing replication-incompetent virus encoding the anti-hCD70 CAR.
* All patients will receive a non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine.
* On day 0, patients will receive PBL transduced with the anti-hCD70 CAR and will then begin high-dose aldesleukin.
* A complete evaluation of lesions will be conducted approximately 6 weeks (plus or minus two weeks) after treatment.
* The study will be conducted using a Phase I/II optimal design, with two separate cohorts for the Phase II component:Cohort 2a, patients with CD70-expressing clear cell renal cell carcinoma (RCC), and Cohort 2b, patients with a CD70-expressing non-RCC malignancy (solid tumors only).
* A total of up to 124 patients may be required; approximately 38 patients in the Phase I portion of the study and 43 (41, plus an allowance of up to 2 non-evaluable) patients in each cohort of the Phase II portion of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For Phase I: Evaluable, unresectable cancer expressing CD70 as assessed by immunohistochemistry of resected tissue (greater than or equal to 2+ CD70 positive on greater than or equal to 50% of cancer cells, or greater than or equal to 1+ CD70 positive on greater than or equal to 75% of cancer cells).
* For Phase II: Measurable (per RECIST v1.1 criteria), unresectable cancer expressing CD70 as assessed by immunohistochemistry of resected tissue (greater than or equal to 2+ CD70 positive on greater than or equal to 50% of cancer cells, or greater than or equal to 1+ CD70 positive on greater than or equal to 75% of cancer cells).
* Confirmation of the diagnosis of cancer by the NCI Laboratory of Pathology.
* Patients must have previously received at least one standard therapy for their cancer (if available) and have been either non-responders (progressive disease) or have recurred.
* Patients with 3 or fewer brain metastases that are less than or equal to 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Age greater than or equal to 18 years and less than or equal to 72 years.
* Clinical performance status of ECOG 0 or 1
* Patients of both sexes must be willing to practice birth control from the time of enrollment on this study and for 12 months after the last dose of combined chemotherapy for women and for four months after treatment for men.
* Women of child-bearing potential must be willing to undergo a pregnancy test prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.

NOTE: Certain malignancies may secrete hormones that produce false positive pregnancy tests. Serial blood testing (e.g. HCG measurements) and/ or ultrasound may be performed for clarification.

-Serology

--Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus be less responsive to the experimental

treatment and more susceptible to its toxicities.)

* Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

  -Hematology
* ANC greater than 1000/mm(3) without the support of filgrastim
* WBC greater than or equal to 2500/mm(3)
* Platelet count greater than or equal to 80,000/mm(3)
* Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.

  -Chemistry
* Serum ALT/AST less than or equal to 5.0 times ULN
* Serum creatinine less than or equal to 1.6 mg/dL
* Total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dL.

  * Patients must have completed any prior systemic therapy at the time of enrollment.

Note: Patients may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to grade 1 or less.

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Subjects must be co-enrolled on the NCI-SB cell harvest protocol 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols).

EXCLUSION CRITERIA:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Concurrent systemic steroid therapy.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* History of hematopoietic autoimmune disease or any autoimmune disease requiring immunosuppressive measures.
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune-competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* For select patients with a clinical history prompting cardiac evaluation: last known LVEF less than or equal to 45%.
* For select patients with a clinical history prompting pulmonary evaluation: known FEV1 less than or equal to 50% predicted.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-related adverse events | From time of cell infusion to two weeks after cell infusion
  Grade and type of toxicity per dose level; fraction of patients who experience a DLT at a given dose level, and number and grade of each type of DLT
Response rate | 6 weeks and 12 weeks following administration of the cell product, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who have a clinical response (PR+CR) to treatment (objective tumor regression)

SECONDARY OUTCOMES:
Frequency and severity of treatment-related adverse events | 6 weeks ( plus or minus 2 weeks) following administration of the cell product
  Aggregate of all adverse events, as well as their frequency and severity

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Diegmann J, Junker K, Gerstmayer B, Bosio A, Hindermann W, Rosenhahn J, von Eggeling F. Identification of CD70 as a diagnostic biomarker for clear cell renal cell carcinoma by gene expression profiling, real-time RT-PCR and immunohistochemistry. Eur J Cancer. 2005 Aug;41(12):1794-801. doi: 10.1016/j.ejca.2005.05.005. PMID 16043348
- [Background] Jilaveanu LB, Sznol J, Aziz SA, Duchen D, Kluger HM, Camp RL. CD70 expression patterns in renal cell carcinoma. Hum Pathol. 2012 Sep;43(9):1394-9. doi: 10.1016/j.humpath.2011.10.014. Epub 2012 Mar 7. PMID 22401771
- [Background] Bowman MR, Crimmins MA, Yetz-Aldape J, Kriz R, Kelleher K, Herrmann S. The cloning of CD70 and its identification as the ligand for CD27. J Immunol. 1994 Feb 15;152(4):1756-61. PMID 8120384
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0131.html